CLINICAL TRIAL: NCT06896396
Title: Icaritin Soft Capsules and TACE Combined with Immunotherapy and Targeted Therapy Versus TACE Combined with Immunotherapy and Targeted Therapy for Unresectable Hepatocellular Carcinoma：a Prospective, Double-arm, Exploratory Study
Brief Title: Icaritin Soft Capsules+TACE+Immunotherapy+Targeted Therapy Versus TACE+Immunotherapy+Targeted Therapy for Unresectable Hepatocellular Carcinoma
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Zhiyong Huang (Other)
Responsible Party: Sponsor-Investigator, Zhiyong Huang, Professor, Tongji Hospital
Organization: Tongji Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: uHCC-AKLD-TJ01
Record Dates: First submitted 2025-03-20; First posted 2025-03-26 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Unresectable Hepatocellular Carcinoma
MeSH Terms: interventions — lenvatinib; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Icaritin soft capsules+TACE+Immunotherapy+Targeted Therapy (Experimental): Icaritin soft capsules，lenvatinib and pabilizumab were started 3-5 days after the first TACE treatment
  Interventions: Drug: Lenvatinib, Pembrolizumab; Drug: Icaritin soft capsules; Procedure: TACE
- TACE+Immunotherapy+Targeted Therapy (Active Comparator): lenvatinib and pabilizumab were started 3-5 days after the first TACE treatment
  Interventions: Drug: Lenvatinib, Pembrolizumab; Procedure: TACE

INTERVENTIONS:
Drug: Lenvatinib, Pembrolizumab — Pabilizumab: intravenously every three weeks Lenvatinib, with a dosage based on body weight: 8 mg (≤60 kg) or 12 mg (>60 kg), once daily
Drug: Icaritin soft capsules — Starting 3-5 days after the first TACE treatment, take 6 capsules orally, twice a day, and swallow them with warm water within 30 minutes after breakfast and dinner
  Arms: Icaritin soft capsules+TACE+Immunotherapy+Targeted Therapy
Procedure: TACE — TACE treatment is strictly in accordance with the Chinese guidelines for clinical practice of transcatheter arterial chemoembolization (TACE) for hepatocellular carcinoma (2023 Edition).

SUMMARY:
Hepatocellular carcinoma (HCC) is one of the most common malignant tumors and the leading cause of cancer-related death worldwide. Surgical resection has always been the best hope for long-term survival of patients with HCC. However, only a few patients have the opportunity to undergo surgery, and more than 70% of HCC patients have lost the opportunity of surgery at the time of diagnosis. The treatment measures for these patients are mainly transcatheter arterial chemoembolization and systemic therapy. In recent years, systemic therapies represented by targeted therapy and immunotherapy have made important progress in the field of liver cancer, improving the survival of patients with advanced unresectable HCC. Icaritin soft capsule is a monomer compound extracted, isolated, purified and enzymatically hydrolyzed from the natural medicinal plant Epimedium. It was approved for marketing on January 10, 2022 for patients with advanced first-line HCC. Icaritin soft capsules have the potential to delay TKI resistance and enhance the efficacy of PD-1 inhibitors. The aim of this study is to explore whetherIcaritin soft capsules and TACE combined with Immunotherapy and Targeted Therapy can improve the therapeutic effect of advanced HCC, ultimately prolong the survival time of patients, and provide a new treatment direction for patients with advanced HCC.

ELIGIBILITY:
Inclusion Criteria:

* 1) Age range: 18-75 years old; 2) Patients diagnosed with hepatocellular carcinoma or cirrhosis through histology/cytology meet the clinical diagnostic criteria for hepatocellular carcinoma by the American Association for the Study of the Liver (AASLD). The clinical diagnostic criteria refer to the "Guidelines for Diagnosis and Treatment of Primary Liver Cancer (2024 Edition)"; 3) Advanced primary liver cancer patients who have not received systematic treatment in the past or advanced liver cancer patients who have not received systematic treatment and have relapsed after radical resection; 4) Diseases are not suitable for radical surgery, transplantation, or ablation, but diseases are suitable for TACE treatment 5) At least one measurable lesion. Single tumor, diameter ≤ 10.0cm or multiple tumors; Number ≤ 10; The tumor burden of the lesion is less than 50%; 6) ECOG score 0-1 points; 7) Child Pugh liver function grade A; 8) Expected lifespan ≥ 3 months; 9) Blood, liver, and kidney function meet the following criteria:

  1. Absolute neutrophil count ≥ 1.0 × 109/L;
  2. Platelet count ≥ 75 × 109/L;
  3. Hemoglobin concentration ≥ 90g/L;
  4. Serum albumin concentration ≥ 28g/L;
  5. Serum total bilirubin ≤ 3 x upper limit of normal (ULN);
  6. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 5 × ULN;
  7. The prothrombin time extension shall not exceed ULN6s;
  8. Creatinine<1.5 × ULN or creatinine clearance rate (CrCl)>60 mL/min (Cockcroft Gault formula); 10) If the patient is HBsAg positive, HBV-DNA should be below 2000 IU/ml (10000 copies/ml) during treatment; 11) Women with fertility must undergo a negative pregnancy test; 12) Acceptable contraceptive methods must be used during the research period; 13) Can understand and be willing to sign a written informed consent form; 14) Capable of swallowing and absorbing oral pills; 15) Use up to 3 types of antihypertensive drugs to fully control blood pressure, defined as systolic/diastolic blood pressure ≤ 150/90 mmHg during screening, and no change in antihypertensive treatment within the first week/week prior to the first cycle.

Exclusion Criteria:

* 1) Diffuse infiltrative lesions of the liver and brain metastases; 2) There are TACE contraindications, such as portosystemic shunt, hepatic blood flow and obvious atherosclerosis; 3) Individuals allergic to intravenous contrast agents; 4) Local treatment has been performed on existing lesions (e.g.: TACE、 Melting, particles TARE、 Hepatic artery infusion chemotherapy or radiotherapy); 5) The subject is unable to undergo enhanced liver CT or MRI scans; 6) Previous history of liver transplantation or current candidate for liver transplantation; 7) Pregnant, lactating women or participants planning to undergo contraceptive procedures within 2 years; 8) Patients with combined HIV and syphilis infections; 9) Patients with other concurrent malignant tumors or other malignant tumors within the first 5 years of enrollment; 10) Patients with severe functional impairments of the heart, kidneys, and other organs; 11) Severe clinical active infection>Level 2 (NCI-CTC version 5.0); 12) Mental illness patients who may affect the informed consent process; The patient is unable to take oral medication; The patient participated in clinical trials of other drugs within 12 months prior to enrollment.

  13) Patients who have experienced esophageal or gastric variceal rupture bleeding within the past 3 months, or have unconfirmed severe varices and are at high risk; 14) Has bleeding or thrombotic disease or is undergoing thrombolytic therapy; 15) Clinical significant hemoptysis or tumor bleeding for any reason within 2 weeks prior to the first administration of the study intervention; 16) Major cardiovascular damage within the 12 months prior to the first administration of the investigational drug, such as a history of NYHA class II or higher congestive heart failure, unstable angina, myocardial infarction or cerebrovascular accident stroke, or arrhythmia related to hemodynamic instability; 17) There is clinically significant ascites during physical examination, which cannot be controlled with medication; 18) History of autoimmune diseases or immunodeficiency, including but not limited to myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, antiphospholipid antibody syndrome, Wegener's granulomatosis, Sjogren's syndrome, Guillain Barr é syndrome, or multiple sclerosis 19) Idiopathic pulmonary fibrosis, organizing pneumonia (such as bronchiolitis obliterans), drug-induced pneumonia, or history of idiopathic pneumonia, or evidence of active pneumonia on chest CT scan during screening 20) Known to be allergic to any component of the investigational drug formulation; 21) Other situations where the researcher deems it inappropriate to participate in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2027-06-01 (Estimated); Study Completion 2028-02-01 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | 12 month
  PFS refers to the time from subject enrollment to disease progression according the Response Evaluation Criteria in Solid Tumors version 1.1 (RECISTv1.1) or death

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | 6 weeks after the first TACE surgery
  ORR refers to the proportion of patients whose tumors shrink to a certain amount and maintain for a certain period of time (6 weeks after first dose of Durvalumab), including CR+PR cases. CR (complete response): disappearance of all target lesions, PR (partial response): reduction of the sum of the length and diameter of the baseline lesions by ≥30%.
Overall Survival (OS) | 18 months
  OS was defined as time from diagnosis to death from any cause or the last follow-up
Duration of Response（DOR） | 18 months
  It refers to the time from the first evaluation of the tumor as CR or PR to the first evaluation as PD or death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: huang zhiyong, Principal Investigator — Tongji Hospital
Locations (1):
- Tongji Hospital, Wuhan, Hubei, China